CLINICAL TRIAL: NCT02676154
Title: A Phase II, Open-Label Exploratory Study Investigating the Efficacy of Toviaz for Treatment of Adult Patients With Spinal Cord Injury With Neurogenic Detrusor Overactivity for Amelioration of Autonomic Dysreflexia(PIIR-AK-TOVIAZ-AD)
Brief Title: Fesoterodine for Amelioration of Autonomic Dysreflexia (AD) Following Spinal Cord Injury (SCI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Pfizer (Industry); International Collaboration on Repair Discoveries (Other); Vancouver Coastal Health (Other Government)
Responsible Party: Principal Investigator, Andrei Krassioukov, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H15-02364; WI207218 (Other Grant/Funding Number: Pfizer Canada Inc)
Record Dates: First submitted 2016-01-27; First posted 2016-02-08 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Autonomic Dysreflexia
Keywords: Episodic Hypertension; Spinal Cord Injury; Traumatic Spinal Cord Injury; Blood Pressure; Fesoterodine; Neurogenic Detrusor Overactivity; Autonomic Dysreflexia; Urodynamic Studies; 24 Hour Ambulatory Blood Pressure Monitoring; Cerebral Blood Flow
MeSH Terms: conditions — Autonomic Dysreflexia; Spinal Cord Injuries | interventions — fesoterodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fesoterodine (Other): Open-Label
  Interventions: Drug: Fesoterodine

INTERVENTIONS:
Drug: Fesoterodine — 4mg, oral, once daily for 12 weeks; dose adjustments may be permitted.
  Other Names: Toviaz

SUMMARY:
This study will be investigating the effects of fesoterodine on autonomic dysreflexia (AD) in patients with spinal cord injuries (SCI). The goal of the study is to examine the effect of increasing daily use of fesoterodine on episodes of high blood pressure triggered by urinary bladder contractions.

DETAILED DESCRIPTION:
This is a Phase 2, open-label exploratory study investigating the efficacy of fesoterodine for treatment of adult patients with spinal cord injuries (SCI) with autonomic dysreflexia (AD) triggered by neurogenic detrusor overactivity (NDO).

ELIGIBILITY:
The inclusion criteria include, but are not limited to, the following:

* Male or female, 18 - 60 years of age
* Chronic traumatic SCI at or above T6 spinal segment and >1 year post injury
* Documented presence of AD and NDO during UDS
* Hand function sufficient to perform CIC or a committed caregiver to provide CIC for management of urinary bladder drainage
* Patients must have documented two weeks of bladder and bowel history prior to their baseline visit
* Willing and able to comply with all clinic visits and study-related procedures
* Able to understand and complete study-related questionnaires (must be able to understand and speak English or have access to an appropriate interpreter as judged by the investigator).
* Women of childbearing potential must not be intended to become pregnant, currently pregnant, or lactating. The following conditions apply:
* Women of childbearing potential must have a confirmed negative pregnancy test prior to the baseline visit. During the trial, all women of childbearing potential will undergo urine pregnancy tests at their monthly clinic visits as outlined in the schedule of events.
* Women of childbearign potential must agree to use adequate contraception during the period of the trial and for at least 28 days after completion of treatment. Effective contraception includes abstinence.
* Sexually active males with female partners of childbearing potential must agree to use effective contraception during the period of the trial and for at least 28 days after completion of treatment
* Must Provide Informed Consent

The exclusion criteria include, but are not limited to, the following:

* Presence of severe acute medical issue that in the investigator's judgement would adversely affect the patient's participation in the study
* A hypersensitivity to tolterodine (available as Detrol, Detrol LA), soya, peanuts, or lactose
* Recent treatment with intravesical OnabotulinumtoxinA (within 9 months of the baseline visit)
* Recent treatment with other anticholinergics medications (within 3 weeks of the baseline visit)
* Use of any medication or treatment that in the opinion of the investigator indicates that it is not in the best interest of the patient to participate in this study
* Patient is a member of the investigational team or his /her immediate family

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Number of participants that experience a decrease in severity of autonomic dysreflexia (AD) from baseline following 12-weeks of study medication. | 12 weeks
Number of participants that experience a decrease in the severity of spontaneously occurring episode of Autonomic Dysreflexia (AD) during the 24 hour Ambulatory Blood Pressure Monitoring (24hr ABPM) | 12 weeks

SECONDARY OUTCOMES:
Number of participants that experience a decrease in the frequency of autonomic dysreflexia (AD) episodes from baseline following 12-weeks of study medication. | 12 weeks
Number of participants that experience an improvement from baseline of self-reported severity and frequency of AD as reported with the Autonomic Dysreflexia Health Related-Quality of Life (AD HR-QoL) questionnaire and reflected by a decrease in score. | 12 weeks
An improvement from baseline of self-reported bladder incontinence as reported with the Incontinence Quality of Life (I-QoL) questionnaire and reflected with an increase in score. | 12 weeks
An improvement from baseline of cognitive function as evaluated with the Montreal Cognitive Assessment scale (MoCA) and reflected with a total score at or greater than 26. | 12 weeks
An improvement from baseline in bowel stool outcomes as reported with the Bristol Stool Scale. | 12 weeks
An Improvement from baseline in the ability of the bladder to stretch in response to filling of the bladder as indicated by Urodynamics Study (UDS) parameters of bladder volume and pressure on the detrusor muscle.. | 12 weeks
An improvement from baseline in Cerebral Blood Flow (CBF) during Urodynamics Study (UDS) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Krassioukov, MD,PhD,FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Data collected during the study will be used by the investigator to communicate results of the study to the research community. Data will mostly be communicated as a pooled data set; in the event that individual participant data is communicated, it will be represented with the unique study identifier which does not identify the individual participant.

REFERENCES:
- [Derived] Walter M, Ramirez AL, Lee AH, Rapoport D, Kavanagh A, Krassioukov AV. Protocol for a phase II, open-label exploratory study investigating the efficacy of fesoterodine for treatment of adult patients with spinal cord injury suffering from neurogenic detrusor overactivity for amelioration of autonomic dysreflexia. BMJ Open. 2018 Nov 21;8(11):e024084. doi: 10.1136/bmjopen-2018-024084. PMID 30467135